CLINICAL TRIAL: NCT04503928
Title: Euphorbia Kansui in Combination With Antiretroviral Therapy for Eradication of the Latent HIV-1 Reservoir
Brief Title: Euphorbia Kansui and HIV/AIDS Functional Cure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: Fudan University (Other); Shanghai Xinhao Biological Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Euphorbia kansui V1
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: All participants eligible for study received the same open label drug
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Kansui 1g per day x 7 days (Experimental): Study participants will be given 1 g of Euphorbia kansui Pill for a total of 7 consecutive daily doses.
  Interventions: Drug: Euphorbia kansui Pill

INTERVENTIONS:
Drug: Euphorbia kansui Pill — 1 g (10 pills) of Euphorbia kansui Pill taken by mouth, once a day for 7 consecutive days.
  Other Names: kansui

SUMMARY:
The purpose of this study is to determine the safety and bioactivity of Euphorbia kansui, which has been used in traditional Chinese medicine for the treatment of edema, ascites, and asthma. The investigators previously reported that effective fractions from the dichloromethane extracts of the roots of Euphorbia kansui can reactivate latent HIV-1 replication in different latent cells (The 24th China science technology Forum-High level Forum on HIV cure, December 16-17, 2012, Beijing). Importantly, in resting CD4+ T cells of HIV-1-infected patients on suppressive antiretroviral therapy (ART), it could effectively induce ex vivo latent HIV-1 expression. Sera from rats receiving orally administered effective fractions were able to reactivate latent HIV-1. The investigators also found a substantially potent ingenol derivative EK-16A, EK-1A, EK-5A, EK-15A from Euphorbia kansui and proved that it was potent in reversing HIV-1 latency. The investigators' hypothesis is that Euphorbia kansui Pill will be safe and well-tolerated and at the doses administered, increase HIV transcription in latently-infected cells among HIV-infected patients on suppressive antiretroviral therapy.

DETAILED DESCRIPTION:
Every participant will receive oral Euphorbia kansui Pill every day. The dose of Euphorbia kansui will be 1g each time for 7 consecutive days. All participants will keep their antiretroviral therapy during this study.

Each step of this study will last for 21 days, involving 7 study visits (Screening,Day 0, 1, 3, 5, 7, 14, 21) for every participant. At the screening visit, participants will give a medical history and will undergo a physical exam; blood samples will be collected. Participants will undergo pharmacodynamic sampling which will require that blood be collected 12 hours after kansui Pill administration on Day 1, 3, 5,7. If participants agree, their blood samples may be stored for future research.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection
2. Age ≥18 years; Willingness to give written informed consent.
3. Karnofsky performance status >70.
4. Able, willing to adhere to therapy and adherent to ART.
5. Able, willing to comply with time requirements for study visits and evaluations.
6. On potent combination ART for ≥ 18 months prior to study entry.
7. Able to swallow pills without difficulty.
8. HIV-1 RNA values <50 copies/mL for at least 18 months.
9. CD4 cell count ≥ 500 cells/µl at screening.
10. CD4 T cells isolated in vitro and stimulated with kansui, and the kansui activation test is positive.
11. All volunteers must agree not to participate in a conception process.
12. Must have adequate organ function as indicated by the following lab values:

Hematological: Absolute Neutrophil Count (ANC) ≥ 1,500/mcL Platelets ≥ 125,000/mcL Hgb ≥ 12 g/dL Coagulation: Prothrombin Time or International Normalized Ratio (INR) ≤ 1.5x upper limit of normal (ULN) Chemistry: K+ levels Within normal limits Mg++ levels > Lower limits of normal (LLN) but <1.5 x ULN Glucose Screening serum glucose(fasting/non-fasting) below 120 mg/dl.

Renal: Serum creatinine/calculated creatinine clearance* ≤ 1.3 X ULN OR ≥ 60 mL/min for participants with creatinine levels > 1.3 X ULN Hepatic: Serum total bilirubin Total bilirubin < 1.5 times ULN. If total bilirubin is elevated, direct bilirubin will be measured and the participant will be eligible if the direct bilirubin is < 2 X ULN.

Aspartate amino transferase (AST) (SGOT) and Alanine amino transferase (ALT) (SGPT)≤ 2.0 X ULN Lipase <1.6 X ULN Alkaline Phosphatase ≤ 2.5 X ULN.

Exclusion Criteria:

1. Acute HIV-1 infection
2. Received blood transfusions or hematopoetic growth factors within 3 months
3. Receipt of compounds with other latency activators within 1 month.
4. Any significant acute medical illness in the past 8 weeks
5. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood
6. Patient has the following laboratory values within 3 weeks before starting the investigational drug Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN) Serum total bilirubin ≥1.5 ULN Serum creatinine levels ≥1.5 x ULN, or calculated creatinine clearance ≤60 ml/min Platelet count ≤100 x109/L Absolute neutrophil count ≤1.5x109/L Serum potassium, magnesium, phosphorus outside normal limits Total calcium (corrected for serum albumin) or ionized calcium ≤lower normal limits
7. A personal history of clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for Torsades de pointes (e.g. heart failure)
8. History of malignancy or transplantation, including skin cancers or Kaposi sarcoma
9. History of diabetes mellitus
10. Known hypersensitivity to Kansui
11. Pregnancy or breast feeding, or expecting to father children within the projected duration of the study
12. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma HIV-1 RNA concentration | Measured on day 0; 1, 3, 5, 7 (12 hours post administration); 14, 21.
Change in cell-associated HIV-1 RNA | on day 0; 1, 3, 5, 7 (12 hours post administration); 14, 21
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Measured through 21 days after the first administration of kansui Pill

SECONDARY OUTCOMES:
Change in cell-associated total HIV-1 DNA | Measured on day 0, 14, 21

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, M.D., Principal Investigator — Shanghai Public Health Clinical Center; Huanzhang Zhu, M.D., Principal Investigator — Fudan University
Locations (1):
- Shanghai,China, Fudan University, Shanghai, China

REFERENCES:
- [Background] Wang P, Lu P, Qu X, Shen Y, Zeng H, Zhu X, Zhu Y, Li X, Wu H, Xu J, Lu H, Ma Z, Zhu H. Reactivation of HIV-1 from Latency by an Ingenol Derivative from Euphorbia Kansui. Sci Rep. 2017 Aug 25;7(1):9451. doi: 10.1038/s41598-017-07157-0. PMID 28842560
- [Background] Yang H, Li X, Yang X, Lu P, Wang Y, Jiang Z, Pan H, Zhao L, Zhu Y, Khan IU, Shen Y, Lu H, Zhang T, Jiang G, Ma Z, Wu H, Zhu H. Dual effects of the novel ingenol derivatives on the acute and latent HIV-1 infections. Antiviral Res. 2019 Sep;169:104555. doi: 10.1016/j.antiviral.2019.104555. Epub 2019 Jul 9. PMID 31295520
- See also: Related Info — http://csm.im.ac.cn/templates/team/introduction.aspx?nodeid=10&page=ContentPage&contentid=1950